CLINICAL TRIAL: NCT01471444
Title: A Randomized Study of Once Daily Fludarabine-Clofarabine Versus Fludarabine Alone Combined With Intervenous Busulfan Followed by Allogeneic Hemopoietic Stem Cell Transplantation for Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: Fludarabine-IV Busulfan ± Clofarabine and Allogeneic Hematopoietic Stem Cell Transplantation for Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0628; NCI-2012-00038 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-09

CONDITIONS: Disorder Related to Bone Marrow Transplantation; Leukemia; Transplantation Infection
Keywords: Blood And Marrow Transplantation; Leukemia; Allogeneic hematopoietic stem cell transplantation; Acute myeloid leukemia; AML; Myelodysplastic syndrome; MDS; Progression free survival; Rate of engraftment; Toxicity; Relapse rate; Graft-vs-host disease; GvHD; Progression-free survival; PFS; Overall survival; OS; Fludarabine; Fludarabine Phosphate; Fludara; Clofarabine; Clofarex; Clolar; Busulfan; Busulfex; Myleran; Thymoglobulin; ATG; Antithymocyte Globulin; Methotrexate; Tacrolimus; Prograf
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Graft vs Host Disease | interventions — fludarabine; fludarabine phosphate; Clofarabine; Busulfan; thymoglobulin; Antilymphocyte Serum; Bone Marrow Transplantation; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Flu + Bu (Experimental): Fludarabine 40 mg/m2 intravenous (IV) over 1 hour. Busulfan dose calculated to achieve a systemic exposure dose of 6000 µMol-min IV over 3 hours every 24 hours. Both delivered for 4 consecutive days (days -6 to -3). Stem cell transplant Day 0.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Thymoglobulin; Procedure: Stem Cell Infusion; Drug: Tacrolimus; Drug: Methotrexate
- Flu +Clo + Bu (Experimental): Fludarabine 10 mg/m2 over 1 hour. Clofarabine 40 mg/m2 diluted in normal saline to produce a final concentration of 0.4 mg/mL, infused over 1 hour. Busulfan dose calculated to achieve a systemic exposure dose of 6000 µMol-min IV over 3 hours every 24 hours, immediately after Clofarabine. All delivered on 4 consecutive days (days -6 through -3). Stem cell transplant Day 0.
  Interventions: Drug: Fludarabine; Drug: Clofarabine; Drug: Busulfan; Drug: Thymoglobulin; Procedure: Stem Cell Infusion; Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Fludarabine — Flu + Bu Group: 40 mg/m2 by vein on Days -6 through -3.
  Flu +Clo + Bu Group: 10 mg/m2 by vein on Days -6 through -3.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Clofarabine — 30 mg/m2 diluted in normal saline to produce a final concentration of 0.4 mg/mL, and infused on Days -6 through -3.
  Other Names: Clofarex; Clolar
  Arms: Flu +Clo + Bu
Drug: Busulfan — Busulfan systemic exposure dose of 6000 µMol-min in normal saline over three (3) hours by vein every twenty-four (24) hours for four (4) consecutive days (days -6 to -3), starting immediately after the completion of Clofarabine. The dose on day -6 to -3 based on pharmacokinetic analysis of target AUC of 4,000 µMol-min ± 5% for 61-70 years of age (without Pharmacokinetics alternate dose 130 mg/m2).
  Other Names: Busulfex; Myleran
Drug: Thymoglobulin — Both groups who receive a graft from an unrelated donor:
  0.5 mg/kg on day -3, 1.5 mg/kg on day -2 and 2.0 mg/kg on day -1. On day -3, administered after the chemotherapy is complete.
  Other Names: ATG; Antithymocyte Globulin
Procedure: Stem Cell Infusion — Cryopreserved bone marrow or peripheral blood progenitor cells infused on day 0.
  Other Names: Bone marrow transplant
Drug: Tacrolimus — Starting dose: 0.015 mg/kg (ideal body weight) as a 24 hour continuous infusion daily adjusted to achieve a therapeutic level of 5-15 ng/ml. Changed to oral dosing when tolerated and can be tapered off after day +90 if no graft versus host disease (GVHD) present.
  Other Names: Prograf
Drug: Methotrexate — 5 mg/m2 by vein on Days 1, 3, 6 and 11 post transplant.

SUMMARY:
The goal of this clinical research study is to learn if combining busulfan with clofarabine and fludarabine can help control the disease better than the previous standard method (using busulfan and fludarabine alone) in patients with AML or MDS. The safety of this combination therapy will also be studied.

DETAILED DESCRIPTION:
Busulfan is designed to kill cancer cells by binding to DNA (the genetic material of cells), which may cause cancer cells to die. Busulfan is commonly used in stem cell transplantation.

Clofarabine is designed to interfere with the growth and development of cancer cells.

Fludarabine is designed to interfere with the DNA of cancer cells, which may cause the cancer cells to die.

Study Groups:

You will be randomly assigned (as in the toss of a coin) to 1 of 2 study groups.

* Group 1 will receive busulfan, fludarabine, and clofarabine.
* Group 2 will receive busulfan and fludarabine.

Both groups will have a stem cell transplant. The stem cells will be given by vein. The cells will travel to your bone marrow where they are designed to make healthy, new blood cells after several weeks.

For a stem cell transplant, the days before you receive your stem cells are called minus days. The day you receive the stem cells is called Day 0. The days after you receive the stem cells are called plus days.

Study Drug Administration and Procedures:

Both groups will receive a "test" dose of busulfan by vein over about 45 minutes to 1 hour. This low-level test dose of busulfan is to check how fast busulfan is processed by your body and cleared from your blood. This information will determine the amount of busulfan you will receive. You may receive the busulfan test dose as an outpatient during the week before you are admitted to the hospital or as an inpatient 8 days before your stem cell transplant.

About 11 samples of blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points and will also help determine your dose of busulfan. These blood samples will be drawn at various times before you receive busulfan and over the next 11 hours. These blood draws will be repeated again on the first day of high-dose busulfan treatment (Day -6, which is 6 days before the transplant).

A heparin lock line will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for the PK tests to be performed for technical or scheduling reasons, you will receive the standard fixed dose of busulfan.

On Days -6 through -3, you will receive fludarabine by vein over 1 hour, then clofarabine (if you are in Group 1) by vein over 1 hour, then busulfan by vein over 3 hours.

After the transplant, you will receive tacrolimus, methotrexate, or other immunosuppressive (lowering the immune system) drugs in the standard manner to lower the risk of graft-vs-host disease (GvHD), a reaction of the donor's immune cells against the recipient's body.

If you are going to be receiving a transplant from an HLA-nonidentical or unrelated donor, you will also receive antithymocyte globulin (ATG) by vein over 4 hours on the 3 days before the transplant. This drug is designed to further weaken your immune system to reduce the risk of rejecting of the transplant.

You will receive filgrastim as an injection under the skin 1 time a day, starting 1 week after the transplant, until your blood cell levels return to normal. Filgrastim is designed to help with the growth of white blood cells.

While you are in the hospital, you will be checked for any side effects as part of your standard of care. Blood (about 2 teaspoons) will be drawn every day to check for side effects, for routine tests, to check your blood counts, kidney and liver function, and to check for infections.

As part of standard care, you will remain in the hospital for about 3-4 weeks after transplant. After you are released from the hospital, you must remain in the Houston area to be monitored for infections and other transplant side effects until about 3 months after transplant. During this time, you will return to the clinic at least 1 time each week. The following tests and procedures will be performed:

* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Around 14-30 days after the transplant (when the transplant "engrafts", or "takes"), you will have a bone marrow aspirate to check the status of the disease.

Around Day 30, and about 3, 6, and 12 months after the transplant, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn to see how well the transplant has taken.
* You will have a bone marrow aspiration to check the status of the disease. To collect a bone marrow aspiration, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

Length of Study:

You will be taken off study 5 years after the end of treatment. You may be taken off study early if the disease gets worse, if you have any intolerable side effects, of if you are unable to follow study directions.

You should talk to the study doctor if you want to leave the study early. If you are taken off study early, you still may need to return for routine post-transplant follow-up visits, if your transplant doctor decides it is needed.

It may be life-threatening to leave the study after you have begun to receive the study drugs but before you receive the stem cells.

This is an investigational study. Busulfan and fludarabine are both FDA approved and commercially available for the treatment of AML and MDS. Clofarabine is FDA approved for treating other types of cancer, but is being used in AML and MDS for research only. The use of these study drugs together at the dose level used in this study is investigational.

Up to 250 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have one of the following hematologic malignancies: a) Acute myeloid leukemia (AML) any stage and cytogenetic risk-group with the only exception being that patients with AML and favorable cytogenetics (t(8;21, inv 16, or t(15;17) who achieve complete remission with one course of induction chemotherapy are not eligible . Patients with treatment related AML are eligible. b) Myelodysplastic syndromes (MDS) with intermediate or high risk International Prognostic Scoring System score (IPSS scores) or treatment related MDS. Patients with low risk MDS are eligible if they fail to respond to hypomethylating agent therapy such as azacitidine or decitabine.
2. Age 3-70 years old. Eligibility for pediatric patients will be determined in conjunction with an MDACC pediatrician.
3. Performance score of >/= 60 by Karnofsky or PS 0 to 2 (ECOG) (age > 12 years), or Lansky Play-Performance Scale >/= 60 or greater (age <12 years).
4. Negative Beta HCG test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization. Women of child bearing potential must be willing to use an effective contraceptive measure while on study.
5. Adequate major organ system function as demonstrated by: Left ventricular ejection fraction of at least 40%.
6. Pulmonary function test (PFT) demonstrating a diffusion capacity of least 50% predicted. For children </=7 years of age who are unable to perform PFT, oxygen saturation >/=92% on room air by pulse oximetry.
7. Creatinine < 1.5 mg/dL. If question about renal function discuss with study chairman and do 24 hour creatinine clearance (clearance should be >50 ml/min).
8. Bilirubin < to 2.0 x normal (except Gilbert's Syndrome). SGPT (ALT) < 200. No evidence of chronic active hepatitis or cirrhosis.
9. Histocompatible stem cell donor: Patients must have an HLA matched related or unrelated donor (HLA A, B, C and DR) willing to donate for allogeneic hematopoietic transplantation. High resolution allele level typing is required for donors other than genotypically identical siblings.
10. No uncontrolled infection. Protocol PI or designé will be final arbiter if there is uncertainty regarding whether a previous infection is controlled on appropriate (antibiotic) therapy.
11. Patient or patient's legal representative, parent(s) or guardian able to sign informed consent.

Exclusion Criteria:

1. Positive for HIV, HBsAg, HCV or other viral hepatitis or cirrhosis from any cause.
2. Prior allogeneic or autologous stem cell transplant using a myeloablative busulfan or total body radiation containing conditioning regimen defined as busulfan-based using a total dose of >/=12 mg/kg given by mouth or >/=10 mg/kg given IV; or a total-body irradiation (> 4 Gy).
3. Active or prior CNS leukemia, unless in complete remission for at least 3 months.
4. Previous therapeutic XRT to the liver as part of involved-field radiation.
5. History of serious chronic mental disorder or drug-abuse accompanied by documented problems of compliance with therapeutic programs.
6. Lack of care-giver for the early (100-day) post-transplant period.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2011-11-02 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, BS,MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruitment from November 2011 to August 2015 at MD Anderson Cancer Center
Groups:
- Arm A (Flu+Bu): Fludarabine 40 mg/m2 intravenous (IV) over 1 hour. Busulfan dose calculated to achieve a systemic exposure dose of 6000 µMol-min IV for 60 years and younger or 4000 uMol-min IV for 61 years and older over 3 hours every 24 hours. Both delivered for 4 consecutive days (days -6 to -3). Stem cell transplant Day 0.
- Arm B (Flu+Clo+Bu): Fludarabine 10 mg/m2 over 1 hour. Clofarabine 40 mg/m2 diluted in normal saline to produce a final concentration of 0.4 mg/mL, infused over 1 hour. Busulfan dose calculated to achieve a systemic exposure dose of 6000 µMol-min IV for 60 years and younger or 4000 uMol-min IV for 61 years and older over 3 hours every 24 hours, immediately after Clofarabine. All delivered on 4 consecutive days (days -6 through -3). Stem cell transplant Day 0.
Period: Overall Study
Arm/Group | Arm A (Flu+Bu) | Arm B (Flu+Clo+Bu)
Started | 133 | 123
Completed | 130 | 120
Not Completed | 3 | 3
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm B (Flu+Clo+Bu): FlFludarabine 10 mg/m2 over 1 hour. Clofarabine 40 mg/m2 diluted in normal saline to produce a final concentration of 0.4 mg/mL, infused over 1 hour. Busulfan dose calculated to achieve a systemic exposure dose of 6000 µMol-min IV for 60 years and younger or 4000 uMol-min IV for 61 years and older over 3 hours every 24 hours, immediately after Clofarabine. All delivered on 4 consecutive days (days -6 through -3). Stem cell transplant Day 0.
- Total: Total of all reporting groups
Arm/Group | Arm A (Flu+Bu) | Arm B (Flu+Clo+Bu) | Total
Number analyzed (Participants) | 130 | 120 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 105 | 103 | 208
  >=65 years | 25 | 15 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 76 | 65 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 3 | 8
  White | 120 | 114 | 234
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 127 | 119 | 246
  Saudi Arabia | 2 | 1 | 3
  Qatar | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Number of events with progression free survival. (Progression is defined as more than 5% blast in the peripheral blood or bone marrow biopsy.) or expired from treatment related mortality post transplant.
Time Frame: From day of transplant to disease of progression or death of any cause, whichever came first, assessed up to 5 years
Measure: Number; unit: Number of events
Arm/Group | Arm A (Flu+Bu) | Arm B (Flu+Clo+Bu)
Number analyzed (Participants) | 130 | 120
Number of events | 69 | 61

2. Secondary Outcome: Overall Survival (OS) Post Transplant at 1, 3 and 5 Years
Description: Number of participants in the study who are alive and disease free at 1, 3 and 5 years post transplant.
Time Frame: Post transplant after 1, 3 and 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Flu+Bu) | Arm B (Flu+Clo+Bu)
Number analyzed (Participants) | 130 | 120
Participants
  1 Year Post Transplant | 83 | 82
  3 Year Post Transplant | 69 | 69
  5 Year Post Transplant | 64 | 63

3. Secondary Outcome: Number of Participants in the Study Who Are With no Grade 3 or 4 Acute Graft-versus-host Disease at Any Time During the First 100 Days Post Transplant.
Description: Number of participants in the study who are with no Grade 3 or 4 acute graft-versus-host disease at any time during the first 100 days post transplant.
Time Frame: 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Flu+Bu) | Arm B (Flu+Clo+Bu)
Number analyzed (Participants) | 130 | 120
Participants | 125 | 115

4. Secondary Outcome: Number of Participants With Non Relapse Mortality at 100 Day Post Transplant
Description: Number of participants expired from complications other than relapsed disease at 100 day Post Transplant.
Time Frame: 100 day Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Flu+Bu) | Arm B (Flu+Clo+Bu)
Number analyzed (Participants) | 130 | 120
Participants | 3 | 6

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 years.
Arm/Group | Arm A (Flu+Bu) | Arm B (Flu+Clo+Bu)
All-Cause Mortality (participants affected / at risk) | 67/130 | 59/120
Serious Adverse Events (participants affected / at risk) | 25/130 | 39/120
Other Adverse Events (participants affected / at risk) | 123/130 | 120/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Flu+Bu) (N=130) | Arm B (Flu+Clo+Bu) (N=120)
GI GvHD (Gastrointestinal disorders) | 2 | 4
Skin GVHD (Skin and subcutaneous tissue disorders) | 2 | 2
Bacterial Infections (Infections and infestations) | 2 | 9
Viral Infections (Infections and infestations) | 4 | 3
Fungal Infections (Infections and infestations) | 2 | 4
BK virus associated hemorrhagic cystitis (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Diffused alveolar hemorrhage (General disorders) | 2 | 2
Fluid overload (General disorders) | 0 | 1
Transcient secondary graft failure (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Pulmonary embolism (Vascular disorders) | 0 | 2
DIC (Vascular disorders) | 0 | 1
Elevated transminitis (Hepatobiliary disorders) | 1 | 1
Ascites (Hepatobiliary disorders) | 0 | 1
VOD/SOS (Hepatobiliary disorders) | 0 | 1
Liver GvHD (Hepatobiliary disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Poor graft function (Blood and lymphatic system disorders) | 2 | 0
ABO incompatibility (Blood and lymphatic system disorders) | 1 | 0
Hemochromatosis (Investigations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Flu+Bu) (N=130) | Arm B (Flu+Clo+Bu) (N=120)
Infections (Infections and infestations) | 103 | 89
ATG induced fevers (Investigations) | 65 | 41
Allergic reaction to ATG (Immune system disorders) | 2 | 4
Fluid overload (General disorders) | 58 | 54
ABO incompatibility (Blood and lymphatic system disorders) | 4 | 0
GI GvHD (Gastrointestinal disorders) | 18 | 17
Mucositis (Gastrointestinal disorders) | 123 | 115
Upper GI GvHD (Gastrointestinal disorders) | 35 | 40
Renal insufficiency (Renal and urinary disorders) | 28 | 25
Liver GvHD (Hepatobiliary disorders) | 25 | 21
Chronic ocular GvHD (Eye disorders) | 23 | 20
Chronic oral GvHD (Gastrointestinal disorders) | 20 | 19
Chronic lung GvGHD (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Neutropenic fevers (Investigations) | 42 | 47
Cardiomyopathy (Cardiac disorders) | 2 | 0
Dysrhythmia (Cardiac disorders) | 4 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 | 18
Skin GvHD (Skin and subcutaneous tissue disorders) | 71 | 83
Hypertension (Vascular disorders) | 38 | 37
Ascites (Hepatobiliary disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 41 | 51
Nausea (Gastrointestinal disorders) | 123 | 120
Hemorrhagic cystits (Renal and urinary disorders) | 2 | 0
BK virus associated hemorrhagic cystitis (Infections and infestations) | 20 | 27
Elevated transminitis (General disorders) | 106 | 120
PRES (Nervous system disorders) | 1 | 3
Headaches (Nervous system disorders) | 10 | 13
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 11 | 12
ATG induced skin rash (Skin and subcutaneous tissue disorders) | 19 | 8
Rash (Skin and subcutaneous tissue disorders) | 14 | 18
Confusions (Nervous system disorders) | 0 | 9
Fevers (General disorders) | 0 | 17
VOD/SOS (Hepatobiliary disorders) | 0 | 2
autoimmune hemolytic anemia (Investigations) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Pulmonary embolism (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT01471444/Prot_SAP_000.pdf